CLINICAL TRIAL: NCT02503046
Title: Estimation of Pentraxin 3 and Porphyromonas Gingivalis Levels in Patients With Rheumatoid Arthritis and Periodontitis- An Observational Study
Brief Title: Estimation of Pentraxin3 and PGingivalis Levels in Patients With Knee Joint and Gum Diseases
Acronym: EP3PGKG
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.G.Shankar, PG Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: D139206062
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis; Chronic Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pooled plaque sample will be collected and sent for DNA Extraction by PCR for asseessment of levels of PGingivalis.
  5ml of blood to be collected from each subject, centrifuged, to separate the plasma for estimation of Pentraxin3 (Quantikine ELISA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Arthritis with Periodontitis: Patients aged between 30-65 years with 6 positive diagnostic criteria for Rhematoid Arthritis. Patients should have Clinical attachment loss >6mm, and Probing pocket depth>5mm in more than 6 teeth to satisfy criteria for periodontitis.
  5ml of blood to be collected from each patient, centrifuged and plasma extracted used for estimation of Pentraxin3(Quantikine ELISA) Pooled plaque sample taken,DNA extracted by PCR for estimation of P.Gingivalis levels.
  Interventions: Other: Estimation of Pentraxin3; Genetic: Estimation of P.Gingivalis levels
- Periodontitis group: Patients aged between 30-65 years with Periodontal findings being presence of atleast 20 teeth in the mouth .More than 6 teeth with Clinical attachment loss >6mm and Probing pocket depth>5mm to satisfy criteria for periodontitis. 5ml of blood to be collected from each patient, centrifuged and plasma extracted used for estimation of Pentraxin3(Quantikine ELISA).
  Pooled plaque sample taken,DNA extracted by PCR for estimation of P.Gingivalis levels..
  Interventions: Other: Estimation of Pentraxin3; Genetic: Estimation of P.Gingivalis levels
- Healthy Subjects: Subjects aged between 30-65 years with no systemic diseases and periodontitis. 5ml of blood to be collected from each patient, centrifuged and plasma extracted used for estimation of Pentraxin3(Quantikine ELISA).
  Pooled plaque sample taken,DNA extracted by PCR for estimation of P.Gingivalis levels..
  Interventions: Other: Estimation of Pentraxin3; Genetic: Estimation of P.Gingivalis levels

INTERVENTIONS:
Other: Estimation of Pentraxin3 — 5ml of blood to be collected from each subject, centrifuged, to separate the plasma for estimation of Pentraxin3 (Quantikine ELISA)
Genetic: Estimation of P.Gingivalis levels — Pooled plaque sample will be collected and sent for DNA Extraction by PCR for assessment of levels of PGingivalis

SUMMARY:
Periodontitis and Rhematoid arthritis are chronic inflammatory diseases which share common risk factors The purpose of this study is to determine if Pentraxin 3 and Porphyromonas Gingivalis levels play an important role in the progression of both the diseases.

DETAILED DESCRIPTION:
Periodontal disease progression might play a significant role in the severity and outcome of systemic diseases like rheumatoid arthritis. Pentraxin3 is a newly discovered inflammatory biomarker. It is a member of acute phase proteins and it has been observed from previous studies that plasma pentraxin3 levels have increased with increasing severity of cardiac and renal problems.

Porphyromonas gingivalis proteinase is responsible for the epitope development in RF-Fc region These proteinases are important virulence factors which lead to degradation of host tissue. Porphyromonas gingivalis is also a key periodonto pathogen. Thus the aim of this study is to compare the plasma pentraxin3 and p.gingivalis levels in patients with periodontitis and rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

30 Patients with rheumatoid arthritis and periodontitis 30 Patients with Chronic periodontitis only 30 Healthy subjects Patients with six positive diagnostic criteria for RA,morning stiffness,at least three areas of swollen joints,arthritis of hand joints,symmetric arthritis,rheumatoid nodules,serum rheumatoid factor.

For periodontal findings patients aged ≥30yrs,attachment level ≥6mm,at least 20 teeth should present, ≥ 2 sites with pocket depths ≥ 5mm

Exclusion Criteria:

Patients with aggressive periodontitis, Smokers, with gross oral pathology or tumors, with any systemic disorder other than rheumatoid arthritis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total 90 Subjects of whom 30 subjects belong to the Arthritis and Periodontitis group,30 subjects belong to the Periodontitis group and 30 subjects from the healthy group
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Estimation of Plasma Pentraxin 3 levels. | 7 Months
  5ml of blood collected from each subject and centrifuged to separate plasma for estimation of Pentraxin3 levels (Quantikine ELISA)

SECONDARY OUTCOMES:
Estimation of P.Gingivalis levels. | 7 Months
  Pooled plaque samples to be collected and sent for DNA Extraction by PCR to estimate the levels of PGingivalis

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Gittaboyina, PG(Perio), Principal Investigator — Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre; Rekha R Koduganti, MDS(Perio), Study Director — Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre
Locations (1):
- Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartold PM, Marino V, Cantley M, Haynes DR. Effect of Porphyromonas gingivalis-induced inflammation on the development of rheumatoid arthritis. J Clin Periodontol. 2010 May;37(5):405-11. doi: 10.1111/j.1600-051X.2010.01552.x. PMID 20507365
- [Background] Luchetti MM, Piccinini G, Mantovani A, Peri G, Matteucci C, Pomponio G, Fratini M, Fraticelli P, Sambo P, Di Loreto C, Doni A, Introna M, Gabrielli A. Expression and production of the long pentraxin PTX3 in rheumatoid arthritis (RA). Clin Exp Immunol. 2000 Jan;119(1):196-202. doi: 10.1046/j.1365-2249.2000.01110.x. PMID 10606983
- [Background] Mercado FB, Marshall RI, Klestov AC, Bartold PM. Relationship between rheumatoid arthritis and periodontitis. J Periodontol. 2001 Jun;72(6):779-87. doi: 10.1902/jop.2001.72.6.779. PMID 11453241